CLINICAL TRIAL: NCT01062035
Title: Peripheral Blood Telomere Length as a Biomarker of Advanced Colorectal Adenomas
Brief Title: Study of a Screening Blood Test to Determine Patients' Potential Risk of Adenomatous or Advanced Colon Polyps (ACPs)
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Douglas L. Riegert-Johnson, M.D., Mayo Clinic Jacksonville
Other Study IDs: 09-000131
Record Dates: First submitted 2010-02-02; First posted 2010-02-04 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Colonic Polyp
Keywords: Advanced colon polyp; Adenomatous colon polyp; Adenoma, villous colon polyp; Advanced colorectal adenomas; Colonic neoplasms; High grade dysplasia; Telomere blood testing
MeSH Terms: conditions — Colonic Polyps; Adenoma; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The only specimens obtained will be blood for PBL DNA. For all subjects two 10 cc EDTA tubes will be obtained and processed into DNA.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ACP (advanced colon polyp) Group: Between the ages of 50 and 60 years old and have an ACP (advanced colon polyp)
- Control Group: Individuals between the ages of 50 and 60 years old who have had a negative screening colonoscopy.

SUMMARY:
The aim of this study is to develop a blood test to determine which patients are at risk for pre-cancerous colon polyps (ACPs: Advanced Colon Polyps). The telomere length of peripheral blood lymphocytes (PBLs) can be measured from a blood sample. Mechanistic pathways and the investigator's preliminary data support PBL telomere length as a biomarker for ACPs. The long-term goal of this project is to decrease deaths from colon cancer by using a blood test to target colonoscopy for those patients who are at high risk for pre-cancerous polyps.

DETAILED DESCRIPTION:
Telomeres are the repetitive DNA sequences that cap both ends of chromosomes. Shortening of peripheral blood lymphocyte (PBL) telomeres has been associated with renal and other cancers. The investigators' preliminary data shows an association between shorter PBL telomere length and ACPs.

I. Specific Aims

1. Develop a DNA and data repository from individuals with advanced colon polyps (ACPs) and controls
2. Confirm that individuals 50 to 60 years of age with ACPs tend to have shorter peripheral blood lymphocyte (PBL) telomeres than those without ACPs
3. Identify a potential optimal PBL telomere length cut-off to differentiate between individuals with ACPs and those without for evaluation in a larger scale study

The over reaching long term goal is to decrease disease and death from colorectal cancer (CRC) using a biomarker strategy to target colonoscopy to those at higher risk.

ELIGIBILITY:
Inclusion Criteria:

Advanced Colon Polyp Group (ACP):

* Must be 50 to 60 years of age with an advanced colon polyp (ACP: advanced colon polyps are those larger than 10 mm, or a colon polyp with high grade dysplasia, or a colon polyp with villous features.

Control Group (Controls):

* Must be 50 to 60 years of age and have had a negative screening colonoscopy.
* Controls will also have no history of adenomatous colorectal neoplasia.

Exclusion Criteria:

* Subjects under 50 years of age
* Subjects over 60 years of age
* Subjects with colon polyps less than 10 mm in size

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Most subjects will be recruited at the time of a clinic visit in primary care, community internal medicine, executive international physicals, and/or during a pre-colonoscopy visit in the GI Department or GI Laboratory. The ACP subjects will be identified primarily from those referred for ACP removal (EMR) and secondarily from those having screening colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2010-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Telomere length are shorter in individuals with colon polyps. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Douglas L Riegert-Johnson, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Jacksonville, Jacksonville, Florida, United States